CLINICAL TRIAL: NCT07014449
Title: An Open-Label, Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic, and Preliminary Efficacy of WBC100 Capsules in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Clinical Trial of WBC100 Capsule in Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Weben Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WB002
Record Dates: First submitted 2025-05-22; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: AML (Acute Myelogenous Leukemia; Relapsed Acute Myelogenous Leukemia; Refractory Acute Myeloid Leukemia; Hematologic Malignancy; C-Myc; Adult Acute Myeloid Leukemia
Keywords: c-Myc; Molecular glue; Acute Myelogenous Leukemia; Relapsed and Refractory Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hematologic Neoplasms; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WBC100 Capsules (Experimental): Participants will take WBC100 capsules orally once daily in 28-day cycles. This arm includes a dose-escalation phase using an accelerated titration combined with the traditional '3+3' design. After a single-patient observation at 0.5 mg, three patients will be enrolled per cohort at each subsequent dose level (1.0, 1.5, 2.0, 2.5, and 3.0 mg). Treatment will continue until disease progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: WBC100 QD

INTERVENTIONS:
Drug: WBC100 QD — WBC100 will be administered orally as capsules once daily in 28-day cycles. The dose-escalation phase follows an accelerated titration combined with the traditional '3+3' design.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of WBC100 capsules in patients with relapsed or refractory acute myeloid leukemia (R/R AML). The main questions it aims to answer are:

* What is the safety and tolerability profile of WBC100 in R/R AML patients?
* Can WBC100 effectively induce remission in R/R AML patients?

Participants will:

* Take WBC100 capsules orally once daily in 28-day treatment cycles;
* Undergo regular safety assessments, including adverse event monitoring and laboratory tests;
* Provide blood samples for pharmacokinetic (PK) analysis;
* Have their remission status and efficacy evaluated according to the ELN2022 criteria.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed informed consent and compliance with study procedures;
* 2. Male or female participants aged ≥18 years at the time of consent;
* 3. Diagnosis of relapsed or refractory acute myeloid leukemia (R/R AML) according to the 2016 World Health Organization (WHO) classification;
* 4. ECOG PS 0-2;
* 5. Life expectancy ≥3 months;
* 6. Adequate bone marrow reserve and organ function as defined below:

  1. Bone marrow reserve: Peripheral WBC < 25 × 10⁹/L (leukocyte-reducing agents are allowed, with a washout period of at least 5 half-lives prior to study drug administration);
  2. Coagulation: International normalized ratio (INR) ≤ 2;
  3. Hepatic function: Total bilirubin (TBIL) ≤ 1.5 × ULN; ALT and AST ≤ 2.5 × ULN. In cases of hepatic involvement: ALT or AST ≤ 5 × ULN, and TBIL ≤ 3 × ULN;
  4. Renal function: Creatinine clearance ≥60 mL/min (Cockcroft-Gault), or serum creatinine ≤1.5 × ULN;
  5. Cardiac function: Left ventricular ejection fraction (LVEF) ≥50%; QTcF ≤450 ms for males, ≤470 ms for females.
* 7. Female participants of childbearing potential and fertile male participants with partners of childbearing potential must use medically approved contraception during treatment and for 6 months after the final dose.

Exclusion Criteria:

* 1. Known hypersensitivity to WBC100 capsules or any of their excipients;
* 2. Diagnosis of acute promyelocytic leukemia (APL);
* 3. Diagnosis of mixed phenotype acute leukemia, chronic myeloid leukemia in blast crisis, or AML transformed from myelodysplastic syndromes (MDS) or myeloproliferative neoplasms (MPN);
* 4. Subjects with relapse after allogeneic HSCT, grade ≥ 2 acute GVHD, extensive chronic GVHD requiring immunosuppressive therapy, or autologous HSCT within the past 90 days;
* 5. Subjects who have undergone major surgery, have active ulcers, or have unhealed wounds within 28 days prior to the first dose;
* 6. Received other investigational drugs or treatments within 28 days prior to the first administration, or are still within the safety follow-up period of another clinical trial;
* 7. Subjects with a history of severe cardiovascular or cerebrovascular conditions, including but not limited to:

  1. Significant arrhythmias or conduction disorders (e.g., ventricular arrhythmias, Grade II-III AV block);
  2. Thromboembolic events requiring anticoagulation or presence of vena cava filter;
  3. NYHA Class III-IV heart failure;
  4. Poorly controlled hypertension (SBP ≥140 mmHg or DBP ≥90 mmHg despite treatment).
* 8. Evidence of severe or uncontrolled systemic diseases, such as refractory effusions, poorly controlled diabetes, or significant disorders of the psychiatric, neurological, cardiovascular, respiratory, endocrine, gastrointestinal, hepatic, or renal systems;
* 9. History or presence of immunodeficiency, autoimmune disease requiring systemic immunosuppressants, or organ transplantation;
* 10. Congestive heart failure, aortic dissection, stroke (excluding lacunar infarct), unstable angina, myocardial infarction, bypass surgery, or pulmonary embolism within 180 days prior to first dosing;
* 11. Known risk factors for QT prolongation, including congenital long QT syndrome or drug-induced arrhythmia history;
* 12. Positive for syphilis antibodies, HIV, active HBV infection (HBsAg+ or HBcAb+ with HBV DNA ≥1000 IU/mL), or active HCV infection (HCV Ab+ with detectable HCV RNA);
* 13. Active infection requiring systemic treatment, including uncontrolled bacterial, viral, or fungal infections;
* 14. Gastrointestinal conditions preventing oral drug intake or absorption, such as severe vomiting, chronic diarrhea, intestinal stoma, malabsorption, or inability to swallow;
* 15. Use of strong CYP450 inhibitors/inducers that cannot be stopped ≥7 days before dosing;
* 16. Receipt of monoclonal antibodies, ADCs, radiotherapy within 28 days (14 days for localized radiotherapy), cytotoxic chemotherapy, targeted small molecules within 14 days or 5 half-lives, or CAR-T therapy within 100 days;
* 17. Receipt of any live or attenuated vaccines (e.g., influenza, varicella) within 28 days;
* 18. History of other malignancies within 2 years, except adequately treated basal cell carcinoma, carcinoma in situ of cervix or breast, or squamous cell carcinoma of the skin;
* 19. History of psychiatric or neurological disorders that may interfere with protocol compliance;
* 20. Inability to tolerate venous blood draws;
* 21. Pregnant or breastfeeding women, or women with positive serum hCG during screening;
* 22. Any condition deemed by the investigator to make the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicities (DLTs) | During the first treatment cycle (28 days)
  Evaluated according to NCI-CTCAE version 5.0.
Incidence and severity of treatment-emergent adverse events (TEAEs) | From first dose to 28 days after the last dose
  Includes lab abnormalities, physical exam findings, vital signs, and ECG changes.
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) | 28 days
  Based on observed DLTs.

SECONDARY OUTCOMES:
Cmax | 28 days
  Peak plasma concentration after one dose
Tmax | 28 days
  Time to peak plasma concentration after one dose
AUC0-t | 28 days
  Area under the plasma concentration versus time curve after one dose and multiple dose; time range from 0 to last point when plasma concentration is detectable
AUC0-inf | 28 days
  Area under the plasma concentration versus time curve; time range from 0 to infinity
T1/2 | 28 days
  Half-life period
λz | 28 days
  Elimination rate constant
CL/F | 28 days
  Apparent clearance
Vz/F | 28 days
  Apparent volume of distribution
Cmax, ss | 28 days
  Steady peak plasma concentration after multiple dose
Cmin, ss | 28 days
  Steady minimal plasma concentration after multiple dose
Cavg | 28 days
  Steady average plasma concentration after multiple dose
Tmax, ss | 28 days
  Time to steady peak plasma concentration after multiple dose
CLss/F | 28 days
  Steady apparent clearance
Vss/F | 28 days
  Steady apparent volume of distribution
ARCmax | 28 days
  Peak concentration cumulative coefficient
ARAUC | 28 days
  AUC cumulative coefficient
DF | 28 days
  Degree of fluctuation
Duration of response (DOR) | 2 years
  The period from the first evaluation of complete response (CR) or partial response (PR) to the first evaluation of progressive disease (PD) or death of any cause
Event-free survival period (EFS) | 2 years
  EFS, defined as the time from the start of the subject's enrollment to the occurrence of any event (treatment failure/relapse after CR, CRh or CRi/permanent termination of treatment for any reason/death from any cause), whichever occurs first.
Overall survival (OS) | 2 years
  From date of treatment start until the date of death due to any cause.

OTHER OUTCOMES:
Exploratory biological analysis of bone marrow aspirate samples | Cycle 1 (28 days)
  Bone marrow aspirate samples will be collected at each tumor assessment, when feasible, for exploratory biological analyses such as C-Myc protein expression.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China